CLINICAL TRIAL: NCT03672071
Title: Effectivity of Combined Use of Ephedrine and Norepinephrine on Maternal Hemodynamics in Patients Undergoing Cesarean Delivery Under Spinal Anesthesia
Brief Title: Effects of Norepinephrine-ephedrine Combination on Maternal Hemodynamics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Celaleddin Soyalp, Assist. prof., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: cesarean
Record Dates: First submitted 2018-08-04; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Cesarean
Keywords: ephedrine; norepinephrine; maternal hemodynamics; spinal anesthesia
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Intervention Model Description: A randomized prospective controlled study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group E (Other): If a 20% decrease in any parameter compared to their baseline levels is sustained, necessary interventions 5 mg Ephedrine i.v. will be administered to patient will be performed. In the case of hypotension,
  Interventions: Other: Ephedrine, Noradrenaline ,ephedrine+Noradrenaline)
- Group NE (Other): .If a 20% decrease in any parameter compared to their baseline levels is sustained, necessary interventions 5 mg Noradrenaline, i.v. will be administered to patient will be performed. In the case of hypotension,
  Interventions: Other: Ephedrine, Noradrenaline ,ephedrine+Noradrenaline)
- Group N (Other): . If a 20% decrease in parameter compared to their baseline levels is sustained, necessary interventions mg Ephedrine + 2.5 mg Noradrenaline i.v. will be administered to patient will be performed. In the case of hypotension,
  Interventions: Other: Ephedrine, Noradrenaline ,ephedrine+Noradrenaline)

INTERVENTIONS:
Other: Ephedrine, Noradrenaline ,ephedrine+Noradrenaline) — If a 20% decrease in any hemodynamic parameter compared to their baseline levels is sustained, necessary interventions will be performed. In the case of hypotension, for all groups

SUMMARY:
The aim of this study is to investigate the effect of combined use of Ephedrine and Norepinephrine on maternal hemodynamics in patients undergoing cesarean delivery under spinal anesthesia. Secondary aim of the study is to investigate the effect of this combination on neonatal Apgar score and umbilical cord blood gas values.

DETAILED DESCRIPTION:
The study will have a double-blind design and will include 90 patients planned for elective cesarean delivery aged 18-45 years with an ASA score of I-II who will be randomized by sealed tender and will be divided into 3 groups with 30 patients each. The exclusion criteria will be as follows: conversion to general anesthesia, an ASA score of III and IV, emergency surgery, hemodynamic instability, maternal cardiac and pulmonary diseases, placenta previa, placental abruption, intrauterine fetal death, expectancy for a syndromic child, intrauterine growth restriction, preeclampsia, a history of allergy to Ephedrine and Norepinephrine, and neonatal intubation after birth due to respiratory distress or other causes. Each patient will undergo physical examination and laboratory testing one day prior to the procedure. On the same day, each patient will be given information about spinal anesthesia and cesarean delivery under spinal anesthesia, and the patients consenting to participate will be included in the study.

Each patient will undergo preoperative examination 30 min prior to the surgery. After establishing intravenous access, crystalloid fluid 10 cc/kg will be injected. The patient will then be transferred to the operating table. Routine monitorization will be performed and preoperative hemodynamic parameters including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP), and blood oxygen saturation (SpO2) will be recorded for each patient.

Spinal Anesthesia Procedure: After placing the patient in the sitting position and ensuring asepsis and antisepsis, the spinal L3-L4 intercostal space will be palpated and 10 mg 0.05% bupivacaine and 25 microgram fentanyl will be administered using a 25-gauge Quincke needle after viewing the cerebrospinal fluid through the arachnoid space, followed by withdrawal of the needle and administration of pressure dressing. Subsequently, the table will be tilted to the left side by 15 degrees and O2 gas flow will be administered through a nasal cannula at a flow rate of 2 L/min. Following the assessment of dermatomal level, surgical procedure will be initiated.

Throughout the surgical procedure, hemodynamic parameters will be recorded using noninvasive methods every 2 min. If a 20% decrease in any hemodynamic parameter compared to their baseline levels is sustained, necessary interventions will be performed. In the case of hypotension, 5 mg Ephedrine, 5 mg Noradrenaline, and 5 mg Ephedrine + 2.5 mg Noradrenaline i.v. will be administered in Groups E, N, and EN, respectively. On the other hand, surgical details including the total number of vasoactive agent administrations and the length of intervals between administrations, frequency of side effects including nausea, vomiting, discomfort, and headache, Apgar scores at min 1 and 5, umbilical cord blood gas values, duration of surgery, and demographic characteristics (e.g. age, height, weight, parity) will be recorded for each patient and will be used for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Term pregnant patients.

Exclusion Criteria:

* A maternal cardiac diseases
* Pulmonary diseases
* Placenta previa
* Placental abruption
* Intrauterine fetal death
* Expectancy for a syndromic child
* İntrauterine growth restriction
* Preeclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Term pregnant patients
Enrollment: 90 (Estimated)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
systolic arterial blood pressure | during operation
  The maximal aortic pressure following ejection is termed the systolic pressure.Throughout the surgical procedure, it will be recorded using noninvasive methods every 2 minute as mm/Hg
diastolic arterial blood pressure | during operation
  The lowest pressure in the aorta, which occurs just before the ventricle ejects blood into the aorta, is termed the diastolic pressure.Throughout the surgical procedure, it will be recorded using noninvasive methods every 2 minute as mm/Hg

CONTACTS AND LOCATIONS:
Overall Officials: CELALEDDİN SOYALP, Principal Investigator — Yuzuncu Yil University Dursun Odabas Medical School Anesthesiology a nd Reanimation Department, Van, Turkey
Locations (1):
- Celaleddin Soyalp, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided